CLINICAL TRIAL: NCT05078528
Title: Low-cost Mobile Colposcopy and Confocal Imaging for Global Prevention of Cervical Cancer
Brief Title: Low-cost Imaging Technology for Global Prevention of Cervical Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Barretos Cancer Hospital (Other)
Collaborators: William Marsh Rice University (Other); M.D. Anderson Cancer Center (Other); Irmandade Santa Casa de Misericórdia de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 38969820.9.1001.5437
Record Dates: First submitted 2021-10-04; First posted 2021-10-14 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Cervical Intraepithelial Neoplasia
Keywords: image analysis; cancer prevention; cervical intraepithelial neoplasia
MeSH Terms: conditions — Uterine Cervical Dysplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental group - MMC (Experimental): Imaging of study participants will be performed during the colposcopy examination. The mobile colposcope and the confocal imaging probe, together referred to as the Multimodal Mobile Colposcope (MMC), will be used to image and/or record videos the cervix. Cervical biopsies will be performed using biopsy forceps per standard protocols.
  Interventions: Device: Multimodal Mobile Colposcope (MMC)

INTERVENTIONS:
Device: Multimodal Mobile Colposcope (MMC) — Women referred for colposcopy due to abnormal cervical screening or follow-up for a history of dysplasia will be recruited into the experimental group of the study. Imaging of study participants will take place during the colposcopy examination.

SUMMARY:
Cervical cancer remains the first or second leading cause of cancer death among women in many low-and middle-income countries. Cervical cancer prevention programs in low-resource settings are hampered by a lack of personnel with appropriate clinical expertise, lack of pathology services, and lack of associated infrastructure. There is an urgent need for appropriate diagnostic tools to enable accurate screening and diagnosis in low-resource settings. The purpose of this study is to develop and validate a low-cost Multimodal Mobile Colposcope (MMC) for global cervical cancer prevention programs. This new device will combine the imaging capabilities of a mobile colposcope with the microscopic imaging capabilities of a fiber-optic confocal imaging probe.

ELIGIBILITY:
Inclusion Criteria:

* Women >25 years of age;
* Women undergoing colposcopy due to abnormal cervical screening or follow-up for a history of dysplasia;
* Women of childbearing potential must have a negative urine or blood pregnancy test;
* Ability to understand and willingness to provide informed consent by signing specific Informed Consent Document.

Exclusion Criteria:

* Women under 25 years of age;
* Women who have undergone hysterectomy with removal of the cervix;
* Women with known allergy to proflavine or acriflavine;
* Women who are pregnant or nursing at the time of enrollment;
* Incapacitated women or in vulnerable situations or who are not willing to give consent;

Min Age: 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1060 (Estimated)
Dates: Start 2021-09-20 (Actual); Primary Completion 2025-08-03 (Estimated); Study Completion 2025-12-03 (Estimated)

PRIMARY OUTCOMES:
Develop and validate a Multimodal Mobile Colposcope (MMC) | Day 1 - at the colposcopy day
  Image data will be used as a training set to develop and refine image analysis algorithms. Multimodal Mobile Colposcope will be compared with colposcopic impression considering clinical performance (sensitivity, specificity, positive and negative predictive values, and area under the Receiver Operating Characteristic (ROC) curve)

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - Irmandade Santa Casa de Misericórdia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Barretos Cancer Hospital, Barretos, São Paulo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hunt B, Fregnani JHTG, Brenes D, Schwarz RA, Salcedo MP, Possati-Resende JC, Antoniazzi M, de Oliveira Fonseca B, Santana IVV, de Macedo Matsushita G, Castle PE, Schmeler KM, Richards-Kortum R. Cervical lesion assessment using real-time microendoscopy image analysis in Brazil: The CLARA study. Int J Cancer. 2021 Jul 15;149(2):431-441. doi: 10.1002/ijc.33543. Epub 2021 Apr 3. PMID 33811763